CLINICAL TRIAL: NCT00000661
Title: The Pharmacokinetics of Zidovudine and Oxazepam Alone and in Combination in the HIV-Infected Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 124
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 1994-12

CONDITIONS: HIV Infections
Keywords: Oxazepam; Drug Evaluation; Drug Interactions; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Oxazepam; Zidovudine

INTERVENTIONS:
Drug: Oxazepam
Drug: Zidovudine

SUMMARY:
To determine if a pharmacokinetic (blood level) interaction exists between zidovudine (AZT) and oxazepam in the HIV-infected patient. Benzodiazepines (such as oxazepam) are among the most frequently prescribed class of drugs and are commonly used therapeutically for patients with chronic disease. This study is important because of the potential for toxicity resulting from a reaction between AZT and benzodiazepines and the likelihood of frequent use of the combination of these drugs in patients with HIV infection.

DETAILED DESCRIPTION:
Benzodiazepines (such as oxazepam) are among the most frequently prescribed class of drugs and are commonly used therapeutically for patients with chronic disease. This study is important because of the potential for toxicity resulting from a reaction between AZT and benzodiazepines and the likelihood of frequent use of the combination of these drugs in patients with HIV infection.

Patients are studied to determine oral and intravenous AZT and single oral dose oxazepam pharmacokinetics. Patients then take AZT and oxazepam together to determine if interactions between the drugs occur.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Stable prescribed dosage of zidovudine (AZT), = or > 500 mg/day.

Allowed:

* Prophylaxis for Pneumocystis carinii pneumonia (PCP) with aerosolized pentamidine.
* Erythropoietin.

Patients must be:

* HIV positive by ELISA and Western blot.
* Currently taking a stable prescribed dosage of 500 mg/day of zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Allergy to benzodiazepines or a previously documented intolerance to zidovudine (AZT) therapy of = or < 600 mg/day.
* Significant underlying medical condition that could impair continuous participation in study.
* Malabsorption syndrome (3 or more loose stools a day for at least 4 weeks associated with an unintentional weight loss of at least 10 percent of body weight).

Concurrent Medication:

Excluded:

* Oral contraceptives.
* Cytotoxic chemotherapy.
* Ganciclovir.
* Flucytosine.
* Probenecid.
* Opiates.
* Valproic acid.
* Sulfa drugs.
* Sucralfate.
* Dapsone.
* Rifampin.
* Antacids within 2 hours of zidovudine (AZT) dose.
* Isoniazid.
* Ketoconazole.
* Pyrimethamine.
* Clindamycin.
* Aspirin.
* Ibuprofen.
* Investigational drugs not specifically allowed.

Patients with the following are excluded:

* Allergy to benzodiazepines or a previously documented intolerance to zidovudine (AZT) therapy of = or < 600 mg/day.
* Significant underlying medical condition that could impair continuous participation in study.
* Unable to take oral medication reliably.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretroviral agents other than zidovudine (AZT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8

CONTACTS AND LOCATIONS:
Overall Officials: Israelski D, Study Chair; Blaschke T, Study Chair
Locations (1):
- Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California, United States

REFERENCES:
- [Background] Mole LA, Israelski DM, Bubp JL, O'Hanley P, Merigan T, Blaschke T. The pharmacokinetics (PK) of zidovudine (ZDV) and oxazepam (OXA) alone and in combination in the HIV-infected patient (ACTG 124). Int Conf AIDS. 1992 Jul 19-24;8(2):B186 (abstract no PoB 3595)
- [Background] Mole L, Israelski D, Bubp J, O'Hanley P, Merigan T, Blaschke T. Pharmacokinetics of zidovudine alone and in combination with oxazepam in the HIV infected patient. J Acquir Immune Defic Syndr (1988). 1993 Jan;6(1):56-60. PMID 8417175